CLINICAL TRIAL: NCT00807131
Title: Effectiveness of a Pharmaceutical Care Program on Primary Care Patients With Uncontrolled Hypertension- A Brazilian Multicenter RCT
Brief Title: Effectiveness of Pharmaceutical Care on Primary Care Patients With Uncontrolled Hypertension
Acronym: EPHACA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Mauro Silveira de Castro, UFRGS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 402736/2005-2
Record Dates: First submitted 2008-10-31; First posted 2008-12-11 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Hypertension
Keywords: pharmacy care; hypertension; primary care; adherence
MeSH Terms: conditions — Hypertension | interventions — Pharmaceutical Services; Counseling; Prescription Fees

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Patient follow-up
  Interventions: Behavioral: Patient follow-up
- 2 (Experimental): Counseling
  Interventions: Behavioral: Counseling
- 3 (Experimental): Drug dispensing
  Interventions: Behavioral: Drug dispensing
- 4 (Active Comparator): pharmacy usual care
  Interventions: Behavioral: pharmacy usual care

INTERVENTIONS:
Behavioral: Patient follow-up — Dader method, which was developed to provide pharmaceutical care, which consists of seven steps covering the evaluation of services, benefits of interventions, and identification of unexpected occurrences. Its objectives are to improve the patient quality of life.
  Other Names: pharmaceutical care
  Arms: 1
Behavioral: Counseling — The pharmacist proceeds the counseling when the patient comes to the pharmacy to take their medicines.
  Other Names: pharmacist counseling
  Arms: 2
Behavioral: Drug dispensing — The pharmacist gives the drugs to the patient with the minimum of information necessary to guarantee a safe and effective drug intake.
  Other Names: dispensing
  Arms: 3
Behavioral: pharmacy usual care — The patient receives no information about their medicines in the pharmacy, unless he asks for it.
  Other Names: usual care
  Arms: 4

SUMMARY:
This randomized clinical trial is a multicentre study conducted at 4 community-based pharmacies within the Brazilian public health service, which freely distributes standardized medicines. The group coordinator is located at the Universidade Federal do Rio Grande do Sul, a public university at Porto Alegre.

DETAILED DESCRIPTION:
Inclusion and exclusion criteria: Potential hypertensive subjects aged above 18 years and and continuously receiving their medicines from the pharmacy are going to be identified through administrative data sources. They must take at least hydrochlorothiazide, and have no modifications on their hypertensive drug prescription on the last 2 months. Patients who have a serious psychiatric disorder or a severe cognitive impairment, blindness, pregnancy or secondary hypertension will be excluded. To be considered eligible, the patients should have a mean systolic and diastolic blood pressure above 140 mmHg and 90 mmHg at the screening visit if there were no COM morbidities associated, and above 130 mmHg and 80 mmHg for high-risk patients, using the validated Omron Hern-705-CP upper arm automated monitor.

Strategy/process by which participants/centres will be selected and recruited to the trial: Research assistants will invite the potential subjects when they attend the pharmacy to take their medicines or via telephone calls. By this moment, they will confirm eligibility and proceed the BP measures. If eligible for the study, the participant will receive all the trial explanations and the written informed consent will be obtained.

Randomization: The random allocation will be stratified by gender through a computer-generated sequence, individually for each centre. To maintain cancel allocation status, opaque, numbered and sealed envelopes will be adopted.

Interventions: Three different kinds of pharmacist services will be adopted, with growing complexity levels: drug dispensing, counseling and patient follow-up for 8 months. These methods are part of the Brazilian pharmaceutical care agreement, developed on the year of 2002, and will be compared with the pharmacy usual care. Seven pharmacists and 12 students were in charge of the pharmaceutical care program. All of them were trained in a 20 hour-course. Procedures details are written in a manual of operations, willing to standardize the interventions.

Outcomes: The primary outcomes are the BP differences between the one measured at 8-month follow-up and the baseline BP and the adherence, determined by 2 ways: a) measurement of plasma levels of hydrochlorothiazide, measured at the beginning and at the end of the study; b) drugs refill along the 8-months prior the randomization and during the 8-months of the trial. The occurrence of drug-related problems will be evaluated as a secondary outcome.

Blindness: Open-label study. Sample size: The study was design to enroll 304 patients equally distributed within the 4 centers, to provide 80% of statistical power to reject the null hypothesis and an error of 5% (two-tailed). Sampling size was calculated on the basis of a standard deviation of 10 mmHg, powered to detect clinically meaningful differences in mean changes of 5 mmHg between usual care and the intervention arms at 8-months follow-up, considering a 20% of drop-outs. Analyses will be conducted on intention-to-treat basis.

• Statistics: To assess for any differences among the intervention groups, the baseline characteristics will be compared performing Pearson χ2 test for categorical variables and F tests for continuous variables, and Fisher Exact test or Kruskal-Wallis if necessary. For the primary outcomes, the same tests will be applied. Analysis of covariance will be used when necessary.

ELIGIBILITY:
Inclusion Criteria:

* Potential hypertensive subjects aged above 18 years and and continuously receiving their medicines from the pharmacy are going to be identified through administrative data sources.
* They must take at least hydrochlorothiazide, and have no modifications on their hypertensive drug prescription on the last 2 months.
* To be considered eligible, the patients should have a mean systolic and diastolic blood pressure above 140 mmHg and 90 mmHg at the screening visit if there were no COM morbidities associated, and above 130 mmHg and 80 mmHg for high-risk patients.

Exclusion Criteria:

* Patients who have a serious psychiatric disorder or a severe cognitive impairment, blindness, pregnancy or secondary hypertension will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2006-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 8 months

SECONDARY OUTCOMES:
adherence | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Castro, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Mauro Silveira de Castro, Porto Alegre, Rio Grande do Sul, Brazil